CLINICAL TRIAL: NCT05092815
Title: A Single-arm, Open Label, Multicenter Phase II Clinical Study in Rare Diseases to Evaluate Safety, Efficacy and PK of HLX208 for Adult Langerhans Cell Histiocytosis (LCH) and Erdheim-Chester Disease (ECD) With BRAF V600E Mutation
Brief Title: The Efficacy and Safety of HLX208 in Adult Langerhans Cell Histiocytosis (LCH) and Erdheim-Chester Disease (ECD) With BRAF V600E Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-LCH/ECD201
Record Dates: First submitted 2021-09-24; First posted 2021-10-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Langerhans Cell Histiocytosis; Erdheim-Chester Disease; LCH; ECD
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Erdheim-Chester Disease | interventions — CCT239065

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 (Experimental): Participants receive HLX208 450mg bid po
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — HLX208 450mg bid po
  Other Names: BRAF V600E inhibitor

SUMMARY:
The purpose of this study was to assess safety, efficacy and PK in adult Langerhans Cell Histiocytosis (LCH) and Erdheim-Chester Disease (ECD) given HLX208 (BRAF V600E inhibitor).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical study;
2. Aged ≥ 18 years;
3. Confirmed adult patients with LCH and/or ECD with BRAF V600E mutation;
4. At least one measurable lesion as per PERCIST v1.0;
5. Expected survival time ≥ 3 months;
6. ECOG score 0-2;

Exclusion Criteria:

1. Previous treatment with BRAF inhibitors or MEK inhibitors;
2. A history of other malignancies within two years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin, adenocarcinoma in situ of the lung, or tumors that do not require interventional treatment after radical surgery;
3. Severe active infections requiring systemic anti-infective therapy;
4. Other anti-tumor treatments, such as chemotherapy, targeted therapy, or radiation therapy (except palliative radiation therapy), may be given during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 1 year
  Objective response rate(assessed by independent review committee (IRC) based on the PERCIST Version 1.0)

SECONDARY OUTCOMES:
AEs | up to 1 year
  Incidence and severity of adverse events
ORR | up to 1 year
  Objective response rate(assessed by the investigator based on the PERCIST v1.0)
ORR | up to 1 year
  Objective response rate(assessed by IRC and the investigator based on the RECIST v1.1)
DCR | up to 1 year
  Disease control rate (assessed by IRC and the investigator as per PERCIST v1.0 and RECIST v1.1 )
TTR | up to 1 year
  Time to response(assessed by IRC and the investigator as per PERCIST v1.0 and RECIST v1.1)
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 1 year
  Progression-free survival (PFS) (assessed by IRC and the investigator as per PERCIST v1.0 and RECIST v1.1 )
OS | from the date of first dose until the date of death from any cause，assessed up to 1 year
  Overall survival
Cmax | from the date of first dose to 85 days
  Maximum Plasma Concentration
Tmax | from the date of first dose to 85 days
  Time of Maximum Plasma Concentration
AUC | from the date of first dose to 85 days
  Area Under the Curve

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No